CLINICAL TRIAL: NCT05478616
Title: To Investigate the Expression of Endometrium During Window of Implantation Between Natural Cycles and Artificial Cycles
Brief Title: Expression of Endometrium During Window of Implantation
Status: Terminated | Type: Observational
Why Stopped: difficult to recruit patients
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Li-Te Lin, Attending doctor, Department of Obstetrics and Gynecology, Principal Investigator, Assistant professor, Kaohsiung Veterans General Hospital.
Other Study IDs: KSVGH22-CT7-07
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Unrecognized Condition
Keywords: window of implantation; endometrium receptivity; frozen embryo transfer cycles; natural cycles; artificial cycles; hormone replacement therapy cycles

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endometrium during the period of window of implantation will be corrected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Natural cycles: Endometrium will be sampled at the day of LH surge + 7 days.
- Artificial cycles: Endometrium will be sampled at the day of P4 + 5 days.

SUMMARY:
The aim of this study was to investigate the expression of endometrium during window of implantation between natural cycles and artificial cycles.

DETAILED DESCRIPTION:
Due to progress of embryo vitrification in recent years, frozen embryo transfer (FET) of in vitro fertilization (IVF) has already been a world trend. The most used two protocols of FET are natural cycles (NCs) and artificial cycles (ACs). Recent studies showed that IVF outcomes of NCs were superior to ACs. We hypothesized that the result may be because of better endometrial receptivity of NCs compared to ACs. In NCs, no hormonal agents were administrated. Thus, endometrial receptivity was not disturbed by hormone and became better. However, there were few studies to explore the issue. Therefore, the aim of this study was to investigate the expression of endometrium during window of implantation (WOI) between NCs and ACs.

The study will be performed from July 1st, 2022 to December 31th, 2023 in our reproductive center. We plan to enroll 60 infertile women who have underwent IVF cycles and would like to receive endometrial receptivity assay. We divide the participants into two groups, NCs and ACs. In NCs, no hormonal agents will be used. We identify ovulation day via serial hormone data and sample endometrium during WOI (LH surge + 7 days). In ACs, first, estrogen will be given for 10~14 days and then transvaginal sonography will be conducted. When endometrial thickness reaches 8 mm at least, progesterone will be prescribed. Endometrium is sampled during WOI (P4 + 5 days). We will record basic characteristics, infertility history, hormone data, ovarian reserve and endometrial thickness of infertile women in both groups. Endometrial samples will be assessed miRNA, implantation factors, uterine NK cells and T cells in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Age: 30-44 years
* BMI: 18~30 kg/m2
* Implantation failure at least two times

Exclusion Criteria:

* Primary ovarian insufficiency
* Congenital uterine anomaly
* Severe intrauterine adhesion
* Malignancy
* Donor cycle

Ages: 30 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Infertile women aged 30-44 years with implantation failure at least two times
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Expression of endometrium | through study completion, an average of 1.5 year
  miRNA

SECONDARY OUTCOMES:
Implantation factors of endometrium | through study completion, an average of 1.5 year
  HOXA10
Immune cells of endometrium | through study completion, an average of 1.5 year
  Uterine NK cells

CONTACTS AND LOCATIONS:
Overall Officials: Li-Te Lin, Study Director — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Teh WT, McBain J, Rogers P. What is the contribution of embryo-endometrial asynchrony to implantation failure? J Assist Reprod Genet. 2016 Nov;33(11):1419-1430. doi: 10.1007/s10815-016-0773-6. Epub 2016 Aug 1. PMID 27480540
- [Result] Bellver J, Simon C. Implantation failure of endometrial origin: what is new? Curr Opin Obstet Gynecol. 2018 Aug;30(4):229-236. doi: 10.1097/GCO.0000000000000468. PMID 29889670
- [Result] Neves AR, Devesa M, Martinez F, Garcia-Martinez S, Rodriguez I, Polyzos NP, Coroleu B. What is the clinical impact of the endometrial receptivity array in PGT-A and oocyte donation cycles? J Assist Reprod Genet. 2019 Sep;36(9):1901-1908. doi: 10.1007/s10815-019-01535-5. Epub 2019 Jul 27. PMID 31352621
- [Result] Cozzolino M, Diaz-Gimeno P, Pellicer A, Garrido N. Evaluation of the endometrial receptivity assay and the preimplantation genetic test for aneuploidy in overcoming recurrent implantation failure. J Assist Reprod Genet. 2020 Dec;37(12):2989-2997. doi: 10.1007/s10815-020-01948-7. Epub 2020 Sep 24. PMID 32974805
- [Result] Simon C, Gomez C, Cabanillas S, Vladimirov I, Castillon G, Giles J, Boynukalin K, Findikli N, Bahceci M, Ortega I, Vidal C, Funabiki M, Izquierdo A, Lopez L, Portela S, Frantz N, Kulmann M, Taguchi S, Labarta E, Colucci F, Mackens S, Santamaria X, Munoz E, Barrera S, Garcia-Velasco JA, Fernandez M, Ferrando M, Ruiz M, Mol BW, Valbuena D; ERA-RCT Study Consortium Group. A 5-year multicentre randomized controlled trial comparing personalized, frozen and fresh blastocyst transfer in IVF. Reprod Biomed Online. 2020 Sep;41(3):402-415. doi: 10.1016/j.rbmo.2020.06.002. Epub 2020 Jun 15. PMID 32723696
- [Result] Bergin K, Eliner Y, Duvall DW Jr, Roger S, Elguero S, Penzias AS, Sakkas D, Vaughan DA. The use of propensity score matching to assess the benefit of the endometrial receptivity analysis in frozen embryo transfers. Fertil Steril. 2021 Aug;116(2):396-403. doi: 10.1016/j.fertnstert.2021.03.031. Epub 2021 Apr 27. PMID 33926718
- [Result] Riestenberg C, Kroener L, Quinn M, Ching K, Ambartsumyan G. Routine endometrial receptivity array in first embryo transfer cycles does not improve live birth rate. Fertil Steril. 2021 Apr;115(4):1001-1006. doi: 10.1016/j.fertnstert.2020.09.140. Epub 2021 Jan 15. PMID 33461752
- [Result] Rienzi L, Gracia C, Maggiulli R, LaBarbera AR, Kaser DJ, Ubaldi FM, Vanderpoel S, Racowsky C. Oocyte, embryo and blastocyst cryopreservation in ART: systematic review and meta-analysis comparing slow-freezing versus vitrification to produce evidence for the development of global guidance. Hum Reprod Update. 2017 Mar 1;23(2):139-155. doi: 10.1093/humupd/dmw038. PMID 27827818
- [Result] Roque M, Haahr T, Geber S, Esteves SC, Humaidan P. Fresh versus elective frozen embryo transfer in IVF/ICSI cycles: a systematic review and meta-analysis of reproductive outcomes. Hum Reprod Update. 2019 Jan 1;25(1):2-14. doi: 10.1093/humupd/dmy033. PMID 30388233
- [Result] Zaat T, Zagers M, Mol F, Goddijn M, van Wely M, Mastenbroek S. Fresh versus frozen embryo transfers in assisted reproduction. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD011184. doi: 10.1002/14651858.CD011184.pub3. PMID 33539543
- [Result] Mackens S, Santos-Ribeiro S, van de Vijver A, Racca A, Van Landuyt L, Tournaye H, Blockeel C. Frozen embryo transfer: a review on the optimal endometrial preparation and timing. Hum Reprod. 2017 Nov 1;32(11):2234-2242. doi: 10.1093/humrep/dex285. PMID 29025055
- [Result] Shaodi Z, Qiuyuan L, Yisha Y, Cuilian Z. The effect of endometrial thickness on pregnancy outcomes of frozen-thawed embryo transfer cycles which underwent hormone replacement therapy. PLoS One. 2020 Sep 24;15(9):e0239120. doi: 10.1371/journal.pone.0239120. eCollection 2020. PMID 32970718
- [Result] Groenewoud ER, Cantineau AE, Kollen BJ, Macklon NS, Cohlen BJ. What is the optimal means of preparing the endometrium in frozen-thawed embryo transfer cycles? A systematic review and meta-analysis. Hum Reprod Update. 2013 Sep-Oct;19(5):458-70. doi: 10.1093/humupd/dmt030. Epub 2013 Jul 2. PMID 23820515
- [Result] Jing S, Li XF, Zhang S, Gong F, Lu G, Lin G. Increased pregnancy complications following frozen-thawed embryo transfer during an artificial cycle. J Assist Reprod Genet. 2019 May;36(5):925-933. doi: 10.1007/s10815-019-01420-1. Epub 2019 Mar 29. PMID 30924053
- [Result] Liu X, Shi W, Shi J. Natural cycle frozen-thawed embryo transfer in young women with regular menstrual cycles increases the live-birth rates compared with hormone replacement treatment: a retrospective cohort study. Fertil Steril. 2020 Apr;113(4):811-817. doi: 10.1016/j.fertnstert.2019.11.023. Epub 2020 Mar 5. PMID 32147171
- [Result] Melnick AP, Setton R, Stone LD, Pereira N, Xu K, Rosenwaks Z, Spandorfer SD. Replacing single frozen-thawed euploid embryos in a natural cycle in ovulatory women may increase live birth rates compared to medicated cycles in anovulatory women. J Assist Reprod Genet. 2017 Oct;34(10):1325-1331. doi: 10.1007/s10815-017-0983-6. Epub 2017 Jun 24. PMID 28647784
- [Result] Wang A, Murugappan G, Kort J, Westphal L. Hormone replacement versus natural frozen embryo transfer for euploid embryos. Arch Gynecol Obstet. 2019 Oct;300(4):1053-1060. doi: 10.1007/s00404-019-05251-4. Epub 2019 Jul 23. PMID 31338657
- [Result] Del Carmen Nogales M, Cruz M, de Frutos S, Martinez EM, Gaytan M, Ariza M, Bronet F, Garcia-Velasco JA. Association between clinical and IVF laboratory parameters and miscarriage after single euploid embryo transfers. Reprod Biol Endocrinol. 2021 Dec 14;19(1):186. doi: 10.1186/s12958-021-00870-6. PMID 34906128
- [Result] Zanatta A, Rocha AM, Carvalho FM, Pereira RM, Taylor HS, Motta EL, Baracat EC, Serafini PC. The role of the Hoxa10/HOXA10 gene in the etiology of endometriosis and its related infertility: a review. J Assist Reprod Genet. 2010 Dec;27(12):701-10. doi: 10.1007/s10815-010-9471-y. Epub 2010 Sep 7. PMID 20821045
- [Result] Merviel P, Challier JC, Carbillon L, Foidart JM, Uzan S. The role of integrins in human embryo implantation. Fetal Diagn Ther. 2001 Nov-Dec;16(6):364-71. doi: 10.1159/000053942. PMID 11694740
- [Result] Wang W, Sung N, Gilman-Sachs A, Kwak-Kim J. T Helper (Th) Cell Profiles in Pregnancy and Recurrent Pregnancy Losses: Th1/Th2/Th9/Th17/Th22/Tfh Cells. Front Immunol. 2020 Aug 18;11:2025. doi: 10.3389/fimmu.2020.02025. eCollection 2020. PMID 32973809
- [Result] Donoghue JF, Paiva P, Teh WT, Cann LM, Nowell C, Rees H, Bittinger S, Obers V, Bulmer JN, Stern C, McBain J, Rogers PAW. Endometrial uNK cell counts do not predict successful implantation in an IVF population. Hum Reprod. 2019 Dec 1;34(12):2456-2466. doi: 10.1093/humrep/dez194. PMID 31825483